CLINICAL TRIAL: NCT07265726
Title: Exploring the Effectiveness of the Intentionality the Matrix of Healing in Enhancing Oral Health Education Outcomes for Community-dwelling Middle-aged and Older
Brief Title: Oral Health Education for Older Adults: Intentionality in Action
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 25MMHIS120e
Record Dates: First submitted 2025-06-13; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-06

CONDITIONS: Intentionality the Matrix of Healing; Community; Middle-aged and Older Adults; Oral Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Participants in the control group will not receive any intentional interview or expressive arts activity during the 6-week intervention period. They will receive oral health education after the same time interval as the experimental arms, ensuring consistency in outcome measurement.
- Expressive Arts Activities Only (Active Comparator): Participants in this arm will engage only in expressive arts activities over a 6-week period. These activities are designed to foster creative engagement and emotional well-being. After the intervention, participants will receive the same oral health education provided to all groups.
  Interventions: Behavioral: Intentional Interview
- Intentional Interview + Expressive Arts Activities (Experimental): Participants in this arm will receive an intervention combining an intentional interview based on the Intentionality Matrix of Healing framework with expressive arts activities. The intentional interview is designed to guide participants in reflecting on personal health-related intentions, while the expressive arts component facilitates emotional expression and engagement. After the 6-week intervention, all participants will also receive standardized oral health education.
  Interventions: Behavioral: Intentional Interview; Behavioral: Expressive Arts Activities

INTERVENTIONS:
Behavioral: Intentional Interview — Participants in this arm will receive an intervention
  Arms: Expressive Arts Activities Only; Intentional Interview + Expressive Arts Activities
Behavioral: Expressive Arts Activities — Participants in this arm will engage only in expressive arts activities over a 6-week period.
  Arms: Intentional Interview + Expressive Arts Activities

SUMMARY:
After obtaining approval from the Institutional Review Board (IRB), the clinical trial will be registered on a designated trial registration website. Participant recruitment will be conducted online. For individuals who meet the inclusion criteria and express interest, the principal investigator will verbally explain the study protocol, go over the informed consent form, and answer any related questions. Potential participants who meet the inclusion criteria and are willing to participate will be given time to consider their involvement in the study.

Inclusion criteria for this study are:

1. Adults aged 40 and older
2. Ability to hear, speak, and read Chinese, and communicate fluently in Mandarin or Taiwanese.

Exclusion criteria include:

1. Being completely edentulous and not using dentures;
2. Having severe food allergies, renal failure, or dysphagia;
3. Being diagnosed with terminal illness under palliative care, severe mental illness, or cognitive impairment;
4. Having a serious health condition that prevents standing or performing oral self-care behaviors.

Upon receiving verbal agreement from potential participants, the study procedure and the contents of the consent form will be explained again. This is a parallel randomized experimental study, with an estimated sample of 90 middle-aged and older adults recruited from the community through online means. Participants will be randomly assigned to one of three groups:

1. intentional interviews combined with expressive arts activities,
2. expressive arts activities only, or
3. control group.

All three groups will receive oral health education before the intervention and six weeks after the intervention. Questionnaire surveys will be conducted one week and one month post-education to collect data on sarcopenia risk, eating assessment, grit, oral health literacy, and oral self-care behaviors. Statistical analyses will be performed on the collected data.

Participants who fully understand the study and agree to participate will sign an informed consent form. Two copies of the consent form will be prepared-one will be kept by the principal investigator, and a photocopy will be given to the participant for personal recordkeeping. Participants retain the right to decline or withdraw from the study at any time, even after signing the consent form. Their withdrawal will not affect their future rights, benefits, or services, and any previously collected data will be deleted upon request.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 40 years or older (Vlietstra et al., 2024).
2. Ability to hear, speak, and read Chinese, with no communication barriers in Mandarin or Taiwanese.

Exclusion Criteria:

1. Edentulous individuals who do not use dentures.
2. Individuals with severe food allergies, renal failure, or dysphagia.
3. Individuals diagnosed with terminal illness under palliative care, severe psychiatric disorders, or cognitive impairments.
4. Individuals with serious medical conditions that prevent standing or performing oral self-care behaviors.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
sarcopenia risk | baseline, one week after the intervention, and at a one-month follow-up
  This study adopted the SARC-F questionnaire proposed by the Asian Working Group for Sarcopenia (AWGS). The tool consists of five questions aimed at assessing muscle function, including grip strength, endurance, walking ability, ability to stand up from a chair, and fall history in the past six months (Ishida et al., 2020). The first four items are scored based on the responses: no difficulty (0 points), some difficulty (1 point), and a lot of difficulty (2 points). The fifth item, fall history, is scored as follows: 0 falls = 0 points, 1-3 falls = 1 point, and 4 or more falls = 2 points. The total score ranges from 0 to 10, with higher scores indicating a greater risk of sarcopenia. A SARC-F score of 4 or higher suggests a positive result for self-screening, indicating the need for further medical evaluation and appropriate diagnostic and treatment interventions.
  The sensitivity, specificity, and positive/negative likelihood ratios of the SARC-F for predicting sarcopenia and its risk
eating assessment | baseline, one week after the intervention, and at a one-month follow-up
  This study utilized the Eating Assessment Tool-10 (EAT-10), a dysphagia screening tool included in the adult oral health assessment form issued by the Department of Oral Health, Ministry of Health and Welfare. The version used is the Chinese translation by Huang (2023) of the original tool developed by Belafsky et al. (2008). The EAT-10 consists of 10 items that assess self-perceived difficulties related to swallowing, encompassing physical, psychological, and social aspects. Example items include: "Swallowing problems have caused me to lose weight" and "Swallowing interferes with my ability to go out for meals." The scale has demonstrated good reliability and validity, with a Cronbach's alpha coefficient of 0.92. The total score ranges from 0 to 40, with a score of ≥3 indicating the presence of swallowing difficulties. Higher scores reflect a greater risk of oral frailty.
grit | baseline, one week after the intervention, and at a one-month follow-up
  This study adopted the Chinese version of the Grit Scale (Grit-10) developed by Duckworth et al. (2009). The scale consists of 10 items across two main factors: passion (reverse-scored items) and perseverance. Example items include: "I often set a goal but later choose to pursue a different one" (passion, reverse-scored) and "I finish whatever I begin" (perseverance). The scale uses a 5-point Likert rating system, ranging from 1 (not at all like me) to 5 (very much like me).
  Scoring is as follows: each item has a maximum score of 5. Odd-numbered items are reverse scored, and even-numbered items are positively scored. The total score of the odd-numbered items divided by 5 gives the passion subscale score, while the total score of the even-numbered items divided by 5 gives the perseverance subscale score. The sum of all 10 items divided by 10 yields the overall grit score.
  Lin (2019) applied this Chinese version to university students and reported a Cronbach's alpha of 0.84 for the ov
oral health literacy | baseline, one week after the intervention, and at a one-month follow-up
  This study adopted the short-form Health Literacy Dental Scale (HeLD-14) developed by Jones et al. (2015), which has a Cronbach's alpha of 0.87. The scale was translated into Simplified Chinese by Liu et al. (2021) (Chinese version of HeLD, HeLD-C), showing a Cronbach's alpha of 0.92, and was later adapted into a Traditional Chinese version by Cheng (2023). The Traditional Chinese version includes 13 items across seven domains:
  Receptivity (e.g., "I care about my dental or oral health needs"),
  Understanding (e.g., "I can fill out dental-related forms"),
  Support (e.g., "I can bring family members or friends to dental visits"),
  Economic Barriers (e.g., "I can afford the cost of dental or oral health care"),
  Utilization (e.g., "I know how to make a dental appointment"),
  Communication (e.g., "I can obtain alternative oral health opinions from other dentists"), and
  Access to Resources (e.g., "I can follow the dentist's instructions").
  The scale uses a 5-point Likert rating system r
oral self-care behaviors | baseline, one week after the intervention, and at a one-month follow-up
  This study adopted the Oral Self-Care Behavior Scale revised by Cheng (2023), originally developed by Ho, Rita Chang et al. (2019). The scale consists of 10 items; example statements include: "I brush my teeth at least twice a day" and "I always brush my teeth before going to bed at night." A 4-point Likert scale is used, ranging from 1 (not at all) to 4 (completely). The total score ranges from 10 to 40, with higher scores indicating better oral self-care behavior. The Cronbach's alpha ranges from 0.78 to 0.87 (Cheng, 2023), demonstrating good reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanzhi, New Taipei City, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Study Protocol (2025-05-16): https://cdn.clinicaltrials.gov/large-docs/26/NCT07265726/Prot_000.pdf